CLINICAL TRIAL: NCT01651845
Title: Evaluation of a 'Hand-held' Fluorescence Digital Imaging Device for Real-Time Advanced Wound Care Monitoring (JDRTC/UHN)
Acronym: JDRTC/UHN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Principal Investigator, Ralph DaCosta, Principal Investigator, University Health Network, Toronto
Other Study IDs: 12-5003-A
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Wounds; Diabetic Foot Ulcers
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Image Guided Intervention: Standard of care white light visual wound assessment followed by fluorescence image-guided wound assessment

SUMMARY:
We have developed an innovative optical molecular imaging platform (called PRODIGI) based on high-resolution fluorescence and white-light technologies in a hand-held, real-time, high-resolution, non-invasive format. PRODIGI offers a non-contact means of obtaining instantaneous image-based measurements of diagnostically-relevant biological and molecular information of a wound and surrounding skin tissues for the first time and could have significant impact on improving conventional wound care, management, and guidance of intervention.

The investigators hypothesize that real-time imaging of tissue autofluorescence signals emanating from endogenous connective tissue (e.g. collagen) and pathogenic bacteria within complex wounds can be used to determine healing status (i.e., collagen re-modeling and wound closure), detect wound bacterial contamination and/or infection that is occult under standard clinical white light evaluation, and guide intervention during wound care.

DETAILED DESCRIPTION:
The investigators have recently developed an innovative optical molecular imaging platform (called PRODIGI) based on high-resolution fluorescence and white-light technologies in a hand-held, real-time, high-resolution, non-invasive format. PRODIGI offers a non-contact means of obtaining instantaneous image-based measurements of diagnostically-relevant biological and molecular information of a wound and surrounding skin tissues for the first time and could have significant impact on improving conventional wound care, management, and guidance of intervention.

In preliminary preclinical testing, the investigators have discovered that when wounds are illuminated by violet/blue light, endogenous collagen in the connective tissue matrix emit a characteristic green fluorescent signal, while most pathogenic bacterial species emit a unique red fluorescence signal due to the production of endogenous porphyrins. Therefore, with autofluorescence imaging, no exogenous contrast agents are needed during imaging, making this approach particularly appealing as a diagnostic imaging method for clinical use.

Based on extensive preclinical studies in our labs, PRODIGI has demonstrated its capability at collecting autofluorescence images of wounds and detecting the presence and relative changes in connective tissue (e.g. collagen) content and bio-distribution involved in wound healing. It can also detect the presence and relative amounts of commensal and pathogenic bacteria within the wound based on autofluorescence alone (these bacteria are invisible to standard visualization with the naked eye using white light), thus providing a measure of infection status. This could significantly impact clinical wound care and management by i) reducing the complications associated with missed detection of bacterial infection under conventional practice, ii) facilitating image-guided wound sampling by targeted swabbing/biopsy and iii) monitoring wound healing and treatment response over time.

Previous Related Studies: A pilot-level clinical study (UHN REB protocol # 09-0015-A, PI: DaCosta, 50 patients imaged to date) performed by our group from 2008-2011 to assess the clinical utility of the device successfully demonstrated that tissue autofluorescence produced by endogenous collagen/elastin in the skin appears green in the fluorescent images, while most clinically-relevant bacterial colonies present in the wound produce a red fluorescence signal caused by endogenous porphyrins. Some bacterial species (e.g. pseudomonas aeruginosa) produce a green fluorescence signal that can be differentiated spectrally and texturally from the fluorescence of the dermis (another hue of green, discernable by our proprietary image analysis software). The PRODIGI device is sensitive enough to detect these green and red fluorescence signals from tissue and bacteria confirming the utility of this compact and portable imaging platform for clinical wound care.

The investigators hypothesize that real-time imaging of tissue autofluorescence signals emanating from endogenous connective tissue (e.g. collagen) and pathogenic bacteria within complex wounds can be used to determine healing status (i.e., collagen re-modeling and wound closure), detect wound bacterial contamination and/or infection that is occult under standard clinical white light evaluation, and guide intervention during wound care.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. males and females
3. new patient to the JDRTC to ensure consistent work-up procedures (as described below) prior to treatment
4. presenting with acute or chronic wounds (i.e., diabetic ulcers or other), with known or unknown infection status.

Exclusion Criteria:

1. treatment with an investigational drug within 1 month before study enrolment
2. any contra-indication to routine wound care and/or monitoring
3. inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at the Judy Dan Research and Treatment Centre in Toronto. Patients of the JDRTC typically present with diabetic foot ulcers. Eighty new patients with wounds will be entered into this trial, based on statistical power-based calculations for sample size determined in collaboration with the UHN Biostatistics Group (assuming one wound per patient).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate effectiveness of the UHN handheld PRODIGI™ imaging device for real-time and non-invasive detection and tracking of pathogenic bacterial presence, contamination and infectious status in complex wounds over time. | After study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ralph S DaCosta, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Judy Dan Research and Treatment Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DaCosta RS, Kulbatski I, Lindvere-Teene L, Starr D, Blackmore K, Silver JI, Opoku J, Wu YC, Medeiros PJ, Xu W, Xu L, Wilson BC, Rosen C, Linden R. Point-of-care autofluorescence imaging for real-time sampling and treatment guidance of bioburden in chronic wounds: first-in-human results. PLoS One. 2015 Mar 19;10(3):e0116623. doi: 10.1371/journal.pone.0116623. eCollection 2015. PMID 25790480